CLINICAL TRIAL: NCT05849467
Title: Central Nervous System Uptake of Anti-CD8+ T Cell Minibodies in Multiple Sclerosis and Progressive Multifocal Leukoencephalopathy: A Pilot Study
Brief Title: Central Nervous System Uptake of Anti-CD8+ T Cell Minibodies in Multiple Sclerosis and Progressive Multifocal Leukoencephalopathy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10001519; 001519-N
Record Dates: First submitted 2023-05-08; First posted 2023-05-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01-15

CONDITIONS: Multiple Sclerosis; Progressive Multifocal Leukoencephalopathy
Keywords: 89 Zr-Df-crefmirlimab; PET Imaging
MeSH Terms: conditions — Multiple Sclerosis; Leukoencephalopathy, Progressive Multifocal

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Multiple Sclerosis (Experimental): MS cohort- Up to four study visits. (1) Baseline; (2) Day 0: MRI brain/spinal cord (with gadolinium) followed by an intravenous injection of anti-CD8 minibody (aka"PET/CT tracer"); (3) Day 1: PET/CT scan(4) Optional Visit: PET/CT scan
  Interventions: Drug: 89 Zr-Df-crefmirlimab
- Other Neuroinflammatory diseases with BBB leakage (Experimental): Up to four study visits: (1) Baseline; (2) Day 0: MRI brain/spinal cord (with gadolinium) followed by an intravenous injection of anti-CD8 minibody (aka "PET/CT tracer"); (3) Day 1: PET/CT scan(4) Optional Visit: PET/CT scan
  Interventions: Drug: 89 Zr-Df-crefmirlimab
- Progressive Multifocal Leukoencephalopathy (Experimental): PML cohort- Up to five study visits. (1) Baseline; (2) Day 0: MRI brain (with gadolinium) followed by an intravenous injection of anti-CD8 minibody (aka "PET/CT tracer"); (3) Day 1: PET/CT scan; (4) Study visit 4 (optional; time-period between study visit 3 and 4 is variable): MRI brain (with gadolinium) followed by an intravenous injection of anti-CD8 minibody (aka "PET/CT tracer") following clinical, radiological and/or laboratory-defined immune reconstitution (spontaneous or facilitated); (5) Study visit 5: PET/ CT scan
  Interventions: Drug: 89 Zr-Df-crefmirlimab

INTERVENTIONS:
Drug: 89 Zr-Df-crefmirlimab — an 80 kDa minibody (Mb) with high
  affinity to CD8 glycoprotein (binding EC50 = 0.4 nM) that is conjugated with deferoxamine (Df)
  and radiolabeled with the positron emitting radionuclide, Zr-89 (T1/2 78.4 hours).

SUMMARY:
Background:

Multiple sclerosis (MS) and progressive multifocal leukoencephalopathy (PML) are disorders that affect the central nervous system (CNS). The CNS includes the brain, spinal cord, and optic nerves. Both diseases can cause muscle weakness and impair vision, speech, and coordination. Researchers are working to better understand how MS and PML affect the CNS.

Objective: To test whether an experimental radioactive tracer (minibody) can help positron emission tomography (PET) scans detect certain immune cells in the CNS of people with MS and PML.

Eligibility:

People aged 18 years and older with MS, other neuroinflammatory diseases with BBB leakage, or PML.

Design:

Participants will come to the clinic for at least 3 visits over 4 to 6 weeks.

Participants will undergo testing. They will have a physical and neurological exam. They will have blood tests and tests of their heart function. They will have a magnetic resonance imaging (MRI) scan of the brain. They may have a spinal tap: Their lower back will be numbed, and a needle will be inserted between the bones of the spine to withdraw fluid from around the spinal cord.

Minibody is given through a tube with a needle placed in a vein in the arm. This takes 5 to 10 minutes. Participants will have heart function tests before and after receiving the minibody.

Participants may have a PET scan on the day of the Minibody and will return the next day for another PET scan. They will lie on a table that moves through a doughnut-shaped machine. This scan will take about 1 hour.

Participants with PML may opt to repeat the minibody infusion and the PET scan within 6 months.

DETAILED DESCRIPTION:
Study Description:

This study will obtain pilot data for noninvasive positron emission tomography (PET) imaging of CD8 plus T lymphocytes in two inflammatory central nervous system (CNS) demyelinating diseases, multiple sclerosis (MS) and progressive multifocal leukoencephalopathy (PML), and other neuroinflammatory diseases by characterizing CNS uptake of anti-CD8 plus T cell antibody fragment (aka minibody ) (89Zr-Df-crefmirlimab), an investigational, intravenous PET tracer.

Objectives:

Primary Objective: To detect and localize infiltration of CD8 plus T cells in the CNS of adults with MS and PML via PET-CT (computed tomography) scans using a minibody with high affinity for CD8 plus T cells.

Secondary Objectives: (1) To characterize safety and tolerability of 89Zr-Df-crefmirlimab in the participant population. (2) For the PML cohort with longitudinal evaluation, to determine the effects of immune reconstitution, either spontaneous or facilitated, on 89Zr-Dfcrefmirlimab uptake. (3) To determine whether 89Zr-Df-crefmirlimab uptake profile is disease specific for MS and PML.

Endpoints:

Primary Endpoints: Standardized uptake values (SUV) in different tissue types (lesions, white matter, gray matter, meninges, choroid plexus, as determined from coregistered MRI) in each cohort (MS or PML) by region-of-interest (ROI) analysis.

Secondary Endpoints: (1) Frequency and nature of adverse events; (2) For the PML cohort with longitudinal evaluation, changes in SUV over time. (3) Compare patterns of uptake distribution across PML, MS, and other neuroinflammatory diseases with BBB leakage.

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

Multiple Sclerosis Inclusion Criteria

* Enrolled in the NINDS Natural History Study for MS (protocol 89-N-0045)
* Able to understand, and willing to sign, a written, informed consent document.
* Willing to comply with all study procedures and available for the duration of the study.
* Male or female, aged >=18.
* Diagnosis of MS according to the 2017 revision of the McDonald diagnostic criteria48 (in the presence or absence of a clinical relapse).

PML Inclusion Criteria

* Enrolled in the NINDS Natural History Study for PML (protocol 13-N-0017)
* Able to understand and willing to sign a written, informed consent document
* Willing to comply with all study procedures and available for the duration of the study.
* Male or female, aged >=18.
* Diagnosis of definite PML according to 2013 AAN Consensus Criteria49 or PML-IRIS based on clinical, radiological and laboratory evidence.

Patients with Known or Suspected Neuroinflammatory Diseases and Evidence of Open BBB Inclusion Criteria

* Clinical evaluation suggesting an inflammatory disorder of the central nervous system other than MS or PML.
* Recent brain MRI (within 1 month) with gadolinium enhancement indicating open BBB.
* Able to understand and willing to sign a written, informed consent document.
* Willing to comply with all study procedures and available for the duration of the study.
* Male or female, aged >=18.

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Pregnant or lactating.
* Contraindications for MRI gadolinium contrast administration or 3T MRI.
* History of, or current diagnosis with, concomitant medical or clinical conditions that would adversely affect participation in this study.
* Weighs > 350 lb (158 kg; weight limit for the scanner table) or is unable to fit within the MRI or PET imaging gantry.
* Severe claustrophobia unresponsive to oral anxiolytics.
* Has an alkaline phosphatase level greater than 2x ULN (unless known to have non-liver related disorder) OR AST greater than 1.5 x ULN OR ALT greater than 1.5 x ULN.
* Has a total bilirubin >1.5X ULN, unless known to have elevated bilirubin due to nonliver related disorder or Gilbert s.
* Creatinine clearance < 60 mL/min as estimated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI)
* For females of reproductive potential: inability to use highly effective contraception for at least one month prior to screening and during study participation.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Infiltration of CD8+ T cells in the CNS of adults with MS and PML via PET-CT scans using a minibody with high affinity for CD8+ T cells. | Day 1 Study Visit
  To detect and localize infiltration of CD8+ T cells in the CNS of adults with MS and PML via PET-CT scans using a minibody with high affinity for CD8+ T cells.

SECONDARY OUTCOMES:
For the PML cohort with longitudinal evaluation, effects of immune reconstitution, either spontaneous or facilitated, on 89Zr-Dfcrefmirlimab uptake. | up to 6 months after first PET/CT scan
  Comparison of SUV before and after immune reconstitution, either spontaneous or facilitated (for participants with optional follow-up imaging).
Safety of 89Zr-Dfcrefmirlimab in the participants with CNS disease. | At each study visit
  To assess the safety of 89Zr-Dfcrefmirlimab in participants with CNS disease.
To determine whether 89Zr-Df-crefmirlimab uptake profile in MS and PML is disease-specific. | Comparison of pattern of PET uptake distribution and SUV profiles in MS, PML, and other neuroinflammatory diseases with BBB leakage.
  Understand the physiological pattern of 89Zr-Df-crefmirlimab distribution corresponding to normal accumulation of CD8+ T cells.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Reich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001519-N.html